CLINICAL TRIAL: NCT01033175
Title: The Clinical Impact of Anemia of Chronic Disease on Chronic Obstructive Pulmonary Disease Patients
Brief Title: The Impact of Anemia of Chronic Disease on Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Paraskevi Argyropoulou, Professor of Pulmonology, Aristotle University of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 8/22.1.08
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2009-12

CONDITIONS: Anemia; COPD
Keywords: COPD; anemia; exercise; cytokines; erythropoietin
MeSH Terms: conditions — Anemia; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD patients with ACD (Other): In the 1st part of this clinical study the prevalence ACD in COPD subjects will be estimated in a consecutive population of COPD subjects who will visit the hospital's pulmonary clinics as outpatients. During the first visit, subjects will give a detailed medical history and will undergo clinical examination and pulmonary function testing 15 minutes post-bronchodilation. Eligible patients will then undergo peripheral venous blood analysis. The first 30 COPD subjects from the population described above, fulfilling the criteria of ACD will constitute the first arm (group of "cases").ACD is defined by low Hb levels (men: <13 mg/dl, women: <12 mg/dl), no other cause of anemia present, normal or increased serum ferritin and decreased total iron binding capacity.
  Interventions: Procedure: maximal cardiopulmonary exercise testing; Procedure: peripheral blood samples
- COPD patients without ACD (Other): Thirty matched patients with COPD without ACD from the initial cohort will constitute the second arm (the "controls")
  Interventions: Procedure: maximal cardiopulmonary exercise testing; Procedure: peripheral blood samples

INTERVENTIONS:
Procedure: maximal cardiopulmonary exercise testing — Cardiopulmonary exercise testing (CPET) will be performed on a cyclic ergometer with continuous monitoring of a 12-lead electrocardiogram, heart rate and blood pressure. While breathing with a mask, the patients will perform a ramp protocol which includes 2-minutes free pedaling and progressive increase of power by 10, 15 or 20 watts/minute; power size will be selected after considering the patient' s daily activity and parameters of pulmonary function. CPET will be performed until exhaustion, unless the subjects reveal symptoms or signs indicating the exercise should stop (e.g. severe breathlessness).
Procedure: peripheral blood samples — Peripheral venous blood samples will be collected again in the morning after a fasting period of ≥12 hours. After immediate centrifugation, aliquots will be stored at -75˚C until analysis. Inflammatory markers and erythropoietin will be analyzed by flow cytometry and by enzyme-linked immunosorbent assay, using commercially available kits.

SUMMARY:
Hypothesis:

The first part of the study is a survey on the prevalence of anemia of chronic disease (ACD) among COPD patients. The 2nd and 3rd part will test 2 null hypotheses (Ho): 1.serum inflammatory markers and plasma erythropoietin do not differ between COPD patients with and without ACD and 2. exercise capacity does not differ between COPD patients with and without ACD.

Rationale-Aim:

ACD is an immune driven disorder, developing in subjects suffering from chronic inflammatory diseases. COPD is a disorder very likely to be associated to ACD due to its systemic inflammatory dimension. Currently, data on the prevalence of ACD and on the level of inflammatory markers which are implicated in the pathogenesis of ACD in COPD subjects are limited and controversial. Furthermore, there is no data on the effect of ACD on exercise capacity of COPD subjects.

Based to the aforementioned, this study has three goals:

1. to determine the prevalence and the epidemiologic characteristics of ACD in a population of clinical stable COPD patients
2. to investigate whether the levels of serum inflammatory markers and of plasma erythropoietin differ between COPD patients with ACD and without ACD
3. to determine potential differences regarding the aerobic exercise capacity between these two groups, using the cardiopulmonary exercise testing (CPET).

ELIGIBILITY:
Inclusion Criteria:

* 1st part of the study:

  * COPD clinically stable (patients with post-bronchodilation FEV1/FVC <0.7 and no acute exacerbations, hospital admissions or treatment changes in the last 3 months).
  * 2nd and 3rd part:
  * As above.

Exclusion Criteria:

* 1st part of the study:

  * history of asthma,
  * history of respiratory infection in the last 3 months
* 2nd and 3rd part: As above and additionally:

  * history of malignancy or haematologic disorder
  * acute or chronic inflammatory disease
  * systematic or autoimmune disorder
  * thyroid disease
  * liver cirrhosis
  * heart failure (ejection fraction <55%)
  * history of gastrointestinal or other hemorrhage
  * renal failure (GFR<60 ml/min/1.73m2)
  * blood transfusion in the last 4 months
  * administration of cortisone in the last month
  * pregnancy
  * mental impairment
  * medical conditions which are contraindications to exercise testing, such as:
* acute myocardial infarction (in the last 6 months)
* unstable angina
* left main coronary stenosis or its equivalent
* syncope
* symptomatic severe aortic stenosis or other moderate stenotic valvular disease
* uncontrolled arrhythmias causing symptoms
* acute pulmonary embolus or pulmonary infarction
* thrombosis of lower extremities
* suspected dissecting aneurysm
* pulmonary oedema
* room air desaturation at rest <85%
* severe untreated arterial hypertension at rest (>200 mmHg systolic, >120 mmHg diastolic)
* high degree atrioventricular block
* hypertrophic cardiomyopathy and
* orthopedic impairment that compromises exercise performance

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is peak oxygen uptake (VO2 peak, ml/kg/min) during maximal cardiopulmonary exercise testing and whether it differs between patients with ACD and COPD and patients with COPD without ACD. | Within 15 days from enrollment

SECONDARY OUTCOMES:
Serum levels of inflammatory markers | Within 15 days from enrollment
Erythropoietin | Within 15 days from enrollment
MRC dyspnea scale | Within 15 days from enrollment
The rest cardiopulmonary exercise testing parameters | Within 15 days from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi Argyropoulou, MD, Prof, Principal Investigator — Aristotle University Of Thessaloniki
Locations (2):
- Greece (2):
  - Department of Pulmonology, Aristotle University of Thessaloniki, Thessaloniki
  - Respiratory Failure Unit, General Hospital "G. Papanikolaou", Thessaloniki

REFERENCES:
- [Background] Weiss G, Goodnough LT. Anemia of chronic disease. N Engl J Med. 2005 Mar 10;352(10):1011-23. doi: 10.1056/NEJMra041809. No abstract available. PMID 15758012
- [Background] Standards for the diagnosis and care of patients with chronic obstructive pulmonary disease. American Thoracic Society. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 2):S77-121. No abstract available. PMID 7582322
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257